CLINICAL TRIAL: NCT00647348
Title: A Phase II Randomised, Placebo-controlled Clinical Trial of Simvastatin in Patients With Secondary Progressive Multiple Sclerosis.
Brief Title: Investigation of Simvastatin in Secondary Progressive Multiple Sclerosis
Acronym: MS-STAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSTC-001; MREC: 07/Q1602/73 (Other: MREC); 2006-006347-31 (EudraCT Number)
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Results first posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-11

CONDITIONS: Secondary Progressive Multiple Sclerosis
Keywords: Secondary progressive Multiple Sclerosis; Simvastatin; MRI
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Simvastatin

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: over-encapsulation of IMP
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 (Active Comparator): Simvastatin 80mg OD
  Interventions: Drug: Simvastatin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — 80mg simvastatin oral once daily for 24 months
  Arms: 1
Drug: Placebo — Oral placebo tablet once daily for 24 months
  Arms: 2

SUMMARY:
To determine whether simvastatin at a dose of 80mg can reduce the rate of whole brain atrophy, as measured by MRI, over a 2-year time-period when compared to placebo.

DETAILED DESCRIPTION:
The study has now completed see Primary publication:

Effect of high-dose simvastatin on brain atrophy and disability in secondary progressive multiple sclerosis (MS-STAT): a randomised, placebo-controlled, phase 2 trial.

Chataway J, Schuerer N, Alsanousi A, Chan D, MacManus D, Hunter K, Anderson V, Bangham CR, Clegg S, Nielsen C, Fox NC, Wilkie D, Nicholas JM, Calder VL, Greenwood J, Frost C, Nicholas R.

Lancet. 2014 Jun 28;383(9936):2213-21. doi: 10.1016/S0140-6736(13)62242-4.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of multiple sclerosis and at randomisation have entered the secondary progressive stage. Steady progression rather than relapse must be the major cause of increasing disability in the preceding 2 years. Progression can be evident from either an increase of at least one point on the EDSS or clinical documentation of increasing disability.
* EDSS 4.0 - 6.5 inclusive
* Women of childbearing age will be required to use appropriate methods of contraception to avoid the unlikely teratogenic effects of simvastatin.
* Able to give written informed consent
* 18 - 65 years

Exclusion Criteria:

* Unable to give informed consent
* Primary progressive MS
* Those that have experienced a relapse or have been treated with steroids (both i.v. and oral) within 3 months of the screening visit. These patients may undergo a further screening visit once the 3 month window has expired and may be included if no steroid treatment has been administered in the intervening period.
* Patient is already taking or is anticipated to be taking a statin.
* Any medications that unfavourably interact with statins: fibrates, nicotinic acid, cyclosporine, azole anti-fungal preparations, macrolideantibiotics, protease inhibitors, nefazodone, verapamil, amiodarone, large amounts of grapefruit juice or alcohol abuse.
* The use of immunosuppressants (e.g. azathioprine, methotrexate, cyclosporine) or disease modifying treatments (avonex, rebif, betaferon, glatiramer) within the previous 6 months.
* The use of mitoxantrone if treated within the last 12 months.
* If the patient has ever been treated with alemtuzumab.
* If screening levels of alanine aminotransferase (ALT), aspartate aminotransferase (AST) or creatine kinase (CK) are three times the upper limit of normal patients should be excluded.
* Patient unable to tolerate baseline scan or scan not of adequate quality for analysis (e.g. too much movement artefact).
* If a female patient is pregnant or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Chataway, MB BCh, PhD, Principal Investigator — Imperial College London
Locations (3):
- United Kingdom (3):
  - MRI Unit, National Society for Epilepsy, Chesham Lane, Chalfont Saint Peter, Buckinghamshire
  - Charing Cross Hospital, Fulham Palace Road, Hammersmith, London
  - Brighton & Sussex University Hospitals NHS Trust, Eastern Road, Brighton

IPD SHARING:
Plan to Share IPD: Yes
We are still analysing post-hoc data. The International Progressive MS Alliance have access to some of the data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: next 2 years
Access Criteria: via the CI

REFERENCES:
- [Result] Chan D, Binks S, Nicholas JM, Frost C, Cardoso MJ, Ourselin S, Wilkie D, Nicholas R, Chataway J. Effect of high-dose simvastatin on cognitive, neuropsychiatric, and health-related quality-of-life measures in secondary progressive multiple sclerosis: secondary analyses from the MS-STAT randomised, placebo-controlled trial. Lancet Neurol. 2017 Aug;16(8):591-600. doi: 10.1016/S1474-4422(17)30113-8. Epub 2017 Jun 7. PMID 28600189
- [Result] Chataway J, Schuerer N, Alsanousi A, Chan D, MacManus D, Hunter K, Anderson V, Bangham CR, Clegg S, Nielsen C, Fox NC, Wilkie D, Nicholas JM, Calder VL, Greenwood J, Frost C, Nicholas R. Effect of high-dose simvastatin on brain atrophy and disability in secondary progressive multiple sclerosis (MS-STAT): a randomised, placebo-controlled, phase 2 trial. Lancet. 2014 Jun 28;383(9936):2213-21. doi: 10.1016/S0140-6736(13)62242-4. Epub 2014 Mar 19. PMID 24655729
- [Derived] Williams TE, Holdsworth KP, Nicholas JM, Eshaghi A, Katsanouli T, Wellington H, Heslegrave A, Zetterberg H, Frost C, Chataway J. Assessing Neurofilaments as Biomarkers of Neuroprotection in Progressive Multiple Sclerosis: From the MS-STAT Randomized Controlled Trial. Neurol Neuroimmunol Neuroinflamm. 2022 Jan 14;9(2):e1130. doi: 10.1212/NXI.0000000000001130. Print 2022 Mar. PMID 35031587

RESULTS

PARTICIPANT FLOW:
Groups:
- Simvastatin 80mg OD: Simvastatin: 80mg simvastatin oral once daily for 24 months
Period: Overall Study
Arm/Group | Simvastatin 80mg OD | Placebo
Started | 70 | 70
Completed | 67 | 64
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin 80mg OD | Placebo | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 70 | 140
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (7.0) | 51.1 (6.8) | 51.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 48 | 97
  Male | 21 | 22 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 69 | 63 | 132
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Whole Brain Volume
Time Frame: 24 months
Population: 1 participant had a missing data
Measure: Mean (Standard Deviation); unit: percentage of brain volumen change
Arm/Group | Simvastatin 80mg OD | Placebo
Number analyzed (Participants) | 66 | 64
percentage of brain volumen change | 0.288 (0.521) | 0.584 (0.498)
Statistical Analysis 1: Comparison: Simvastatin 80mg OD vs Placebo; Test type: Other — intention-to-treat analysis; p = 0.003, BBSI=brain boundary shift integral

2. Secondary Outcome: Evaluation of Disability (EDSS).
Description: Score (0 to 10), lower score less disability and better progression. For EDSS, mean score at 24 months was compared between treatment groups using an ANCOVA model adjusting for baseline score and minimisation variables.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Simvastatin 80mg OD | Placebo
Number analyzed (Participants) | 67 | 61
score on a scale | 5.93 (1.11) | 6.35 (0.83)
Statistical Analysis 1: Comparison: Simvastatin 80mg OD vs Placebo; Test type: Superiority; p = 0.05, ANCOVA — EDSS,mean score at 24 months was compared between treatment groups using an ANCOVA model adjusting for baseline score and minimisation variables; EDSS,mean score at 24 months was compared between treatment groups using an ANCOVA model adjusting for baseline score and minimisation variables

3. Secondary Outcome: Evaluation of Disability (MSFC Z Score).
Description: Negative value implies worsening and a positive value implies improvement.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Simvastatin 80mg OD | Placebo
Number analyzed (Participants) | 58 | 49
score on a scale | -0.78 (2.06) | -1.21 (2.59)

4. Secondary Outcome: Evaluation of Disability (MSFC Walk).
Description: The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: foot per second
Arm/Group | Simvastatin 80mg OD | Placebo
Number analyzed (Participants) | 62 | 54
foot per second | 1.83 (1.61) | 1.55 (1.19)

5. Secondary Outcome: Evaluation of Disability (MSFC Peg Test).
Description: The patient is seated at a table with a small, shallow container holding nine pegs and a wood or plastic block containing nine empty holes. On a start command when a stopwatch is started, the patient picks up the nine pegs one at a time as quickly as possible, puts them in the nine holes, and, once they are in the holes, removes them again as quickly as possible one at a time, replacing them into the shallow container. The total time to complete the task is recorded.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: speed per second
Arm/Group | Simvastatin 80mg OD | Placebo
Number analyzed (Participants) | 61 | 54
speed per second | 0.033 (0.010) | 0.033 (0.010)

6. Secondary Outcome: Evaluation of Disability (MSFC PASAT).
Description: The PASAT is a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability. Single digits are presented every 3 seconds and the patient must add each new digit to the one immediately prior to it. Shorter inter-stimulus intervals, e.g., 2 seconds or less have also been used with the PASAT but tend to increase the difficulty of the task. Score 0 to 60, higher score less disability.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Simvastatin 80mg OD | Placebo
Number analyzed (Participants) | 61 | 50
score on a scale | 38.3 (15.4) | 35.2 (18.0)

7. Secondary Outcome: Disease Impact Specific to the Disease and Rated by the Patient (MSIS-29 Questionnaire Total Score)
Description: The MSIS-29 is a 29-item self-report measure with 20 items associated with a physical scale and 9 items with a psychological scale. Items ask about the impact of MS on day-to-day life in the past two weeks. All items have 5 response options: 1 "not at all" to 5"extremely". Each of the two scales is scored by summing the responses across items, then converting to a 0-100 scale where 100 indicates a greater impact of the disease on daily function (worse health).
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Simvastatin 80mg OD | Placebo
Number analyzed (Participants) | 66 | 57
score on a scale | 70.1 (15.6) | 76.1 (16.3)

8. Secondary Outcome: Disease Impact Specific to the Disease and Rated by the Patient (MSIS-29 Questionnaire Physical Score)
Description: The MSIS-29 is a 29-item self-report measure with 20 items associated with a physical scale and 9 items with a psychological scale. Items ask about the impact of MS on day-to-day life in the past two weeks. All items have 5 response options: 1 "not at all" to 5"extremely". Each of the two scales are scored by summing the responses across items, then converting to a 0-100 scale where 100 indicates greater impact of disease on daily function (worse health).
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Simvastatin 80mg OD | Placebo
Number analyzed (Participants) | 66 | 57
score on a scale | 51.7 (11.4) | 56.3 (11.8)

9. Secondary Outcome: Disease Impact Specific to the Disease and Rated by the Patient (MSIS-29 Questionnaire Psychological Score)
Description: as for outcome 7
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Simvastatin 80mg OD | Placebo
Number analyzed (Participants) | 66 | 57
score on a scale | 18.3 (5.8) | 19.8 (6.0)

ADVERSE EVENTS:
Time Frame: Collected over 24 months
Arm/Group | Simvastatin 80mg OD | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 9/70 | 14/70
Other Adverse Events (participants affected / at risk) | 49/70 | 54/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simvastatin 80mg OD (N=70) | Placebo (N=70)
Grade 3 relapse (requiring hospital admission) (Immune system disorders) | 3 | 5
Abdominal Lesion Biopsy (Gastrointestinal disorders) | 0 | 1
Appendectomy (Gastrointestinal disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Seizures (Nervous system disorders) | 1 | 0
Increased spasticity (Nervous system disorders) | 0 | 1
Sub-arachnoid haemorrhage (Nervous system disorders) | 0 | 1
Urinary tract infection (Renal and urinary disorders) | 2 | 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Viral encephalitis (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Simvastatin 80mg OD (N=70) | Placebo (N=70)
Relapse (Nervous system disorders) | 17 | 17 — relapse of MS
cramp (Nervous system disorders) | 12 | 10 — cramp
headache (Musculoskeletal and connective tissue disorders) | 3 | 10 — headache
pain (General disorders) | 7 | 13 — pain
worsening mobility (Nervous system disorders) | 9 | 8 — worsening mobility
increase spasticity (Nervous system disorders) | 0 | 7 — spasticity
Urinary infection (Infections and infestations) | 9 | 8 — UTI

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No